CLINICAL TRIAL: NCT04551807
Title: Multi-center, Parallel-group, Randomized Controlled Trial of Modified Natural Versus Programmed Cycles for Frozen Embryo Transfers and Their Association With Preeclampsia and Live Births
Brief Title: Natural Versus Programmed Frozen Embryo Transfer (NatPro)
Acronym: NatPro
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: JHSPH Center for Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00214688
Record Dates: First submitted 2020-08-27; First posted 2020-09-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related; Pre-Eclampsia
Keywords: frozen embryo transfer; infertility; in vitro fertilization
MeSH Terms: conditions — Pre-Eclampsia; Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified natural cycle (Active Comparator): corpus luteum present
  Interventions: Procedure: Modified natural cycle
- Programmed cycle (Active Comparator): corpus luteum absent
  Interventions: Procedure: Programmed cycle

INTERVENTIONS:
Procedure: Modified natural cycle — This treatment protocol is defined as a modified natural cycle as the participant will be instructed to (1) administer human chorionic gonadotropin (hCG) to assist with timing of the embryo transfer and (2) supplement the luteal phase with a low dose of progesterone.
  Arms: Modified natural cycle
Procedure: Programmed cycle — This protocol is designated as programmed because the endometrial development occurs only in association with administration of estradiol and progesterone. No ovulation occurs due to suppression of follicle development by the estradiol and the timing of the transfer is based on the number of days elapsed following initiation of exogenous progesterone.
  Arms: Programmed cycle

SUMMARY:
NatPro is a two-arm, parallel-group, multi-center, randomized trial in which women undergoing frozen embryo transfer (FET) will be randomized to receive either a modified natural cycle (corpus luteum present) or a programmed cycle (corpus luteum absent).

DETAILED DESCRIPTION:
NatPro is a two-arm, parallel-group, multi-center, randomized trial in which women undergoing FET will be randomized to receive either a modified natural cycle (corpus luteum present) or a programmed cycle (corpus luteum absent). The study will implement a stratified randomization design to balance the use of pre-implantation genetic testing (PGT) across the two treatment arms. Each participant will have up to 3 FET cycles until live birth occurs, or the participant has no embryos available for transfer. Primary endpoints will be the proportion of women experiencing preeclampsia comparing modified natural to programmed FET among women with viable pregnancy (defined as pregnancy lasting at least 20 weeks) and the cumulative proportion of women having live births in the two arms.

ELIGIBILITY:
Inclusion criteria

To be eligible, subjects must meet all these criteria:

* Age 18-39 years at the time that embryos were created if no PGT testing was performed. If PGT testing was performed and indicates that an embryo is euploid, the patient can be included if she was age 18-41 years at the time that the embryo was created.
* Age 18-41 years at the time of randomization as advancing age itself becomes a significant risk for preeclampsia
* Normal uterine cavity as assessed by saline infusion sonohysterogram, hysterosalpingogram, or hysteroscopy within one year of the enrollment visit, and repeated at the discretion of the investigator
* Regular menstrual cycle length (approximately 24-35 days) indicative of ovulatory cycles.
* Willing to undergo elective single embryo transfer
* Body Mass Index <=40
* If Body Mass Index is over 30 or individual has other risk factors for diabetes, normal hemoglobin A1C
* Prior to enrollment, participant will have at least one vitrified blastocyst with euploid result by pre-implantation genetic testing (PGT-A) or at least one vitrified blastocyst of fair or better morphologic quality if no PGT-A results are available.
* Willingness to be randomized to either a modified natural or programmed cycle, with a willingness to administer intramuscular progesterone in oil if assigned to the programmed cycle.
* Normal thyroid stimulating hormone (TSH), according to local laboratory standards (or TSH level with a clinically insignificant abnormality per the site director), within one year of study enrollment and repeated at the discretion of the investigator. Use of thyroid medication is permitted.

Exclusion criteria

To be eligible, subjects must not meet any one of these criteria:

* Medical contraindication to pregnancy
* Embryos created using donor oocytes
* Embryo donation
* Gestational carrier
* Reciprocal IVF (one female partner carrying pregnancy, other female partner as source of eggs)
* Fresh embryos created from frozen oocytes. Patients with frozen embryos created from frozen oocytes can be included.
* Recurrent implantation failure defined as no clinical pregnancy with ≥ 2 prior consecutive embryo transfers unless patient also had successful live birth between or after the failed embryo transfers
* Anti-phospholipid antibody syndrome or rheumatologic disease requiring chronic systemic medications
* Uncontrolled diabetes mellitus
* History of >1 pregnancy loss in the second or third trimester
* Uncontrolled hypertension
* Untreated hydrosalpinx (i.e., hydrosalpinx in situ which has not been ligated or removed)
* Mullerian uterine anomaly, if not correctable
* Physician recommendation to perform the embryo transfer outside of the timing specified by the protocol
* Contraindication to any medication which must be used in preparation for the frozen embryo transfer (i.e., estradiol, progesterone, hCG)

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women attempting to get pregnant using frozen embryos
Enrollment: 788 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Preeclampsia | During pregnancy through the post-partum period, according to ACOG guidelines (typically between 20 weeks gestation and 6 weeks post-delivery)
  Frequency of preeclampsia, as defined by American College of Obstetricians and Gynecologists (ACOG) guidelines for hypertensive disorders in pregnancy (Obstetrics & Gynecology 2020;135:e237-e260)

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Baker, MD, Principal Investigator — Department of Gynecology and Obstetrics, Johns Hopkins School of Medicine; James Segars, MD, Principal Investigator — Department of Gynecology and Obstetrics, Johns Hopkins School of Medicine
Locations (15):
- United States (15):
  - University of California San Francisco, San Francisco, California
  - Stanford University, Sunnyvale, California
  - Yale, Orange, Connecticut
  - Fertility Institute of Hawaii, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins, Baltimore, Maryland
  - Shady Grove Fertility, Rockville, Maryland
  - Boston IVF, Waltham, Massachusetts
  - University of Rochester, Rochester, New York
  - Atrium Health, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Beachwood, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - CARE Fertility, Bedford, Texas
  - West Virginia University Center for Reproductive Medicine, Morgantown, West Virginia

REFERENCES:
- [Background] Baksh S, Casper A, Christianson MS, Devine K, Doody KJ, Ehrhardt S, Hansen KR, Lathi RB, Timbo F, Usadi R, Vitek W, Shade DM, Segars J, Baker VL; NatPro Study Group. Natural vs. programmed cycles for frozen embryo transfer: study protocol for an investigator-initiated, randomized, controlled, multicenter clinical trial. Trials. 2021 Sep 27;22(1):660. doi: 10.1186/s13063-021-05637-3. PMID 34579768